CLINICAL TRIAL: NCT05152836
Title: The Effect of Vibrotractile Stimulation on Parkinson's Tremor - an Explorative Study
Brief Title: The Effect of Vibrotactile Stimulation on Parkinson's Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Donders Centre for Cognitive Neuroimaging (Other)
Collaborators: Parkinson's Foundation (Other)
Responsible Party: Principal Investigator, Franziska Goltz, Investigator, Donders Centre for Cognitive Neuroimaging
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL77202.091.21; 2021-12968 (Other: Commissie Mensgebonden Onderzoek)
Record Dates: First submitted 2021-11-25; First posted 2021-12-10 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease; Tremor
Keywords: Parkinson disease; Vibrotactile stimulation; Tremor
MeSH Terms: conditions — Parkinson Disease; Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vibrotactile stimulation atdifferent settings (Experimental): All participants receive vibrotactile stimulation at three different stimulation settings as well as one sham condition. Specifically, stimulation is applied at (1) brief bursts of 80Hz that occur at the individual tremor frequency, (2) 80Hz bursts at tremor frequency*1.5, and (3) continuous stimulation at 80Hz. The sham condition does not involve any stimulation. All of the stimulations will be applied under three different contextual manipulations: during rest, posture and cognitive coactivation (serial subtraction task). Within each context, stimulation/sham conditions are applied in random order.
  Interventions: Device: Vibrotactile stimulation at tremor frequency; Device: Vibrotactile stimulation at tremor frequency*1.5; Device: Vibrotactile stimulation at continuous stimulation; Device: Vibrotactile stimulation 10% below and above step frequency

INTERVENTIONS:
Device: Vibrotactile stimulation at tremor frequency — Mechanical vibrations are applied at brief bursts of 80Hz that occur at the individual tremor frequency. Vibrations are delivered via a small device, which is worn on the wrist of the most-affected arm.
Device: Vibrotactile stimulation at tremor frequency*1.5 — Mechanical vibrations are applied at 80Hz bursts at individual tremor frequency*1.5. Vibrations are delivered via a small device, which is worn on the wrist of the most-affected arm.
Device: Vibrotactile stimulation at continuous stimulation — Continuous 80Hz stimulation is applied via a small device worn on the wrist of the most-affected arm.
Device: Vibrotactile stimulation 10% below and above step frequency — This intervention is applied during assessment of gait. Two devices are worn on both ankles which allows alternating stimulation of both ankles with brief bursts of 80 HZ at the individual step frequency plus or minus 10%.

SUMMARY:
Tremor in Parkinson's disease is a common and highly burdensome symptom. Recent evidence shows that areas in the brain that are underlying Parkinson's tremor overlap with those that respond to somatosensory stimulation. Applying such stimulation to the tremulous limb might therefore influence tremor-related brain activity and thereby potentially reduce tremor. In this study, the investigators explore this possibility and investigate whether tremor specific vibrotactile stimulation at the wrist of the most affected arm influences tremor severity.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disease, of which tremor is a common and highly burdensome symptom. The pathophysiology of tremor involves a cerebral network that consists of basal ganglia and a cerebello-thalamo-cortical motor circuit. Emerging evidence suggests that somatosensory input from the tremulous limb to the brain may influence this network. Specifically, tremor-related activity was observed in primary and secondary somatosensory cortex, and thalamic cells involved in tremor appear to be responsive to somatosensory stimulation as well. Somatosensory afferents may thus play a role in tremor pathophysiology and could therefore be used as treatment target. Here, the investigators will test this hypothesis by investigating the effect of modulating somatosensory input (with vibrotactile stimulation) on tremor severity.

The primary objectives are 1) to test whether rhythmic somatosensory input (vibrotactile stimulation) at tremor frequency reduces tremor power of Parkinson's tremor as compared to vibrotactile stimulation at 1.5 times tremor frequency and 2) whether continuous 80Hz vibrotactile stimulation reduces tremor power as compared to sham stimulation. As secondary objectives, the investigators will test whether the effect of vibrotactile stimulation on tremor power depends on the context in which tremor occurs (rest, cognitive coactivation, posture), whether stimulation at tremor frequency reduces tremor power as compared to sham stimulation, and whether vibrotactile stimulation has an effect on two other common PD symptoms: impaired gait and bradykinesia. The investigators will include 27 patients with Parkinson's disease and rest as well as postural tremor. The intervention involves subtle mechanical vibrations on the wrist or ankles. This is a non-invasive and painless way to provide somatosensory stimuli, in a continuous (80Hz) or rhythmic fashion (brief bursts of 80 Hz at tremor or step frequency).

The investigators expect that this study will provide mechanistic insights into if and how somatosensory (vibro-tactile) afferents influence the cerebral tremor circuit in Parkinson's disease, and may provide a solid basis for designing further clinical treatment studies.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old and able to provide informed consent
* Have a diagnosis of idiopathic PD made by a movement disorders specialist
* Medically optimized without planned medication changes for the duration of the study • Resting tremor subscore >/= 2 of the most-affected arm on the Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) item 2.10
* Postural tremor subscore >/= 1 of the most-affected arm on the MDS-UPDRS item 3.15
* Signed informed consent

Exclusion Criteria:

* The presence of additional neurologic diseases that might confound testing or the coexistence of PD and essential tremor together (action tremor that was present prior to the development of parkinsonism)
* Moderate to severe peripheral neuropathy (reduced vibratory sensation) at the upper extremities, quantified with a graduated tuning fork
* Montreal cognitive assessment (MoCA) score < 20 or previously documented dementia
* Unable to walk without walking aid

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
The effect of vibrotactile stimulation at tremor frequency on tremor severity with active control | 25 minutes
  The investigators will investigate the effect of frequency specific stimulation compared to an active control condition, averaged across three different contexts (rest/posture/cognitive coactivation). Specifically, we will test the change in log transformed tremor power from baseline to stimulation, as a function of stimulation setting (bursts at tremor frequency vs. bursts at 1.5 times tremor frequency).
The effect of continuous vibrotactile stimulation on tremor severity | 25 minutes
  The investigators will investigate the effect of continuous stimulation compared to sham stimulation, averaged across three different contexts (rest/posture/cognitive coactivation). Specifically, we will test the change in log transformed tremor power from baseline to stimulation, as a function of stimulation setting (continuous 80Hz stimulation vs. sham). For the two primary outcomes measures, Bonferroni correction will be applied to correct for multiple comparisons.

SECONDARY OUTCOMES:
The effect of vibrotactile stimulation at tremor frequency on tremor severity with passive control | 25 minutes
  The investigators will explore the change in log transformed tremor power from baseline to stimulation, as a function of stimulation setting (bursts at tremor frequency vs. sham).
The effect of continuous vibrotactile stimulation on bradykinesia | 10 minutes
  The average button presses per second in the keyboard finger tapping test during continuous 80Hz stimulation versus sham will be investigated.
The effect of vibrotactile stimulation on gait | 10 minutes
  Time to complete the timed up and go task will be investigated, comparing stimulation 10% above step frequency/10% below step frequency/sham
The effect of vibrotactile stimulation on freezing | 10 minutes
  Number of freezing episodes during the timed up and go task will be investigated, comparing stimulation 10% above step frequency/10% below step frequency/sham
Investigating the effect of vibrotactile stimulation at tremor frequency on tremor severity in 3 different contexts | 25 minutes
  The investigators will explore the change in log transformed tremor power from baseline to stimulation as a function of stimulation setting (bursts at tremor frequency/bursts at 1.5 times tremor frequency) and context (rest/posture/cognitive coactivation).
Investigating the effect of continuous stimulation on tremor severity in 3 different contexts | 25 minutes
  The investigators will explore the change in log transformed tremor power from baseline to stimulation, as a function of stimulation setting (continuous 80Hz stimulation vs. sham) and context (rest/posture/cognitive coactivation).

CONTACTS AND LOCATIONS:
Overall Officials: Rick C. Helmich, MD PhD, Principal Investigator — Radboud University Nijmegen Medical Centre Donders Institute for Brain, Cognition and Behavior
Locations (1):
- Donders Centre for Cognitive Neuroimaging, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No